CLINICAL TRIAL: NCT06610591
Title: Evaluating the Efficacy of Surgical Intervention for Idiopathic Toe Walking: A Prospective Cohort Pilot Study
Brief Title: Efficacy of Surgery for Idiopathic Toe Walking
Acronym: FOREFOOT
Status: Recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: British Society for Children's Orthopaedic Surgery (Unknown)
Responsible Party: Sponsor
Other Study IDs: PID:17261
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Idiopathic Toe-walking
Keywords: Children; Child; Paediatric; Pediatric; Idiopathic Toe-Walking; Surgery; Orthopaedic; Orthopedic; Pilot; FOREFOOT; Achilles Tendon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Achilles Lengthening Surgery: Participants will receive Achilles lengthening surgery, as usual care.
  Interventions: Procedure: Achilles Lengthening Surgery

INTERVENTIONS:
Procedure: Achilles Lengthening Surgery — The procedure is undertaken under general anaesthetic and involves horizontal hemi-section of the Achilles tendon via small 'stab' incisions at three levels to effect a lengthening of the tendon. The patient is then placed in a walking cast for four weeks thereafter. This surgery is usual care for most children with symptomatic ITW with plantarflexion contractures who have failed non-operative management.

SUMMARY:
BACKGROUND:

For children who walk on their tip toes, surgery is often done to lengthen their Achilles Tendon. However, there is little research to help children's surgeons choose which children with idiopathic toe walking should have surgery.

METHODS:

This research study will investigate how effective surgery to lengthen the Achilles Tendon is for children with idiopathic toe walking. It will explore if the children's quality of life, endurance, strength, range of movement or walking pattern improves after they have had surgery.

This study is a pilot study with 20 participants. This means the results will be used to decide if a larger trial is needed.

DETAILED DESCRIPTION:
BACKGROUND:

It is common for children who learn to walk to walk on their tiptoes to help with their balance. However, approximately 7% of children will continue to walk on their toes past the age of three, with no diagnosis to explain why. This is called as idiopathic toe walking and can cause problems with balance, pain and playing sports.

For children with idiopathic toe walking who cannot touch their heels to the floor in standing, surgery is often done to lengthen their Achilles Tendon. This makes it easier to bend their foot towards their shin. They should then be able to walk. with their heels down in a more typical walking pattern.

However, this improvement is not always long-term. Some children experience problems after surgery, including weak legs. There is little research to help children's surgeons choose which children with idiopathic toe walking should have surgery.

METHODS:

This research study will investigate how effective surgery to lengthen the Achilles Tendon is for children with idiopathic toe walking. It will take part in two hospitals, Oxford University Hospitals and St George's Hospitals. It will explore if the children's quality of life, endurance, strength, range of movement or walking pattern improves after they have had surgery. This study is a pilot study. This means it is a smaller trial with 20 participants. The results will be used to decide if a larger trial is needed, and how a larger trial should be run.

The children in the study will be 8-16 years old, with a tight Achilles Tendon, who have been selected for surgery. They will receive usual care. This means their surgery will be no different than if they were not included in the study.

The children will be given questionnaires with a maximum of 22 questions before surgery, six months after surgery and one year after surgery. They will also do a single heel-rise test before surgery and one year after surgery. This will test if their calf muscle strength has changed after surgery. They will also complete a computerised walking analysis before surgery and one year after surgery. This will test if their walking pattern has changed after surgery. They will also complete a satisfaction questionnaire one year after surgery. This will ask about how satisfied they are with the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 8-16 at recruitment.
* Idiopathic toe walkers based on clinicians' assessment.
* Plantarflexion contracture with knee extended of 0 degrees or less of dorsiflexion.
* Listed for surgical lengthening of the plantarflexors.

Exclusion Criteria:

* Unable to give informed assent or consent. Previous surgery to the lower limb.
* Unable to effectively participate in gait analysis (e.g. unable to walk 10-metres unaided, unable to walk independently, allergy to adhesive for skin markers, hyperhidrosis).
* Underlying diagnoses which may cause toe walking (e.g. muscular dystrophy, split cord malformation, cerebral palsy).
* Listed for additional procedures in the surgery for the lengthening of the plantarflexors.
* Awaiting further investigations or neurology assessment for toe walking pattern.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The population relevant to this study will be children aged 8-16 years old (inclusive) with idiopathic toe walking, estimated to affect 5% of healthy children.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Oxford Ankle Foot Questionnaire for Children (OxAFQ-C) | Pre-surgery / six months post-surgery / one year post-surgery
  Quality of life tool

SECONDARY OUTCOMES:
EuroQol 5 Dimensions Youth (EQ-5D-Y) | Pre-surgery / six months post-surgery / one year post-surgery
  Health related quality of life
Single heel rise test | Pre-surgery / one year post-surgery
  Calf endurance test
Ankle range of motion | Pre-surgery / one year post-surgery
  Measured with a long arm goniometer
Single question | Pre-surgery / six months post-surgery / one year post-surgery
  Thinking of your child's walking over the past week, approximately how much of the time does your child walk on their tiptoes?
Patient Reported Experience Measure (PREM) | One year post-surgery
  Satisfaction with the surgical outcome
Three Dimensional Gait Analysis (3DGA) | Pre-surgery / one year post-surgery
  The comparisons of interest from the 3DGA will be the change from baseline to 1 year, and comparison between participants and age/gender matched control dataset at both time points in:
  Kinetics/Kinematics:
  * Mean pelvic tilt
  * Peak dorsiflexion angle during stance
  * Peak dorsiflexion angle during swing
  * Hindfoot inversion/eversion during stance
  * Peak knee flexion during stance
  * Peak internal plantarflexion moment
  * Peak internal knee flexion moment
  * Peak ankle power generation
  * Gait profile score
  Temporal parameters:
  * Normalised speed (metres per second, normalised for leg length/height)
  * Cadence (steps per minute)
  * Non dimensional stride length (metres, normalised to leg length)

CONTACTS AND LOCATIONS:
Overall Officials: Alpesh Kothari, MA, BM, BCh, AFHEA, MSc, DPhil, Principal Investigator — University of Oxford; Yael Gelfer, BSc, MD, PhD, FRCS, Study Director — St George's University Hospitals NHS Foundation Trust; Julie Stebbins, DPhil SRCS CSci, Study Director — University of Oxford
Locations (2):
- United Kingdom (2):
  - St George's University Hospitals NHS Foundation Trust, Tooting, London
  - Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire

IPD SHARING:
Plan to Share IPD: No
This was not included in the participant information sheets.